CLINICAL TRIAL: NCT06211816
Title: Efficacy of End-of-life Communication Strategies on Nurses in the Intensive Care Unit: A Single-center Before and After Study
Brief Title: Efficacy of End-of-life Communication Strategies on Nurses in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maebashi Red Cross Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 000001
Record Dates: First submitted 2023-12-07; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurse prior to intervention (Other)
  Interventions: Other: communication strategy

INTERVENTIONS:
Other: communication strategy — an intensive communication strategy on end-of-life practice was implemented, based on a framework developed by the International Delphi Conference.

SUMMARY:
Burnout among healthcare workers is frequently reported, and one of the factors cited is the stress caused by end-of-life care. It has been reported that nursing staff experience decreased well-being as a result of being involved in end-of-life care, and this is also true in intensive care units. This decrease in well-being is said to lead to lower quality of care, poor communication with patients and their families, absenteeism, and high turnover. Although palliative care interventions such as education and communication tools have been reported to improve the well-being of healthcare professionals involved in end-of-life care, few reports have evaluated the association with burnout. We investigated whether communication-based palliative interventions in end-of-life care in intensive care units (ICUs) improve the risk of burnout among nurses working in ICUs.

DETAILED DESCRIPTION:
A before-and-after study was conducted in a single hospital to evaluate burnout risk and satisfaction with end-of-life situations in 2022 (phase 1) and 2023 (phase 2). The Japanese version of the Burnout Scale was used to assess the risk of burnout, and the QODD (Quality of Dying and Death) was used to assess nurse satisfaction. All nurses who agreed to participate received the questionnaire in a sealed envelope, completed it, and returned it anonymously to the principal investigator. Data from those who declined to participate were not recorded. During the first and second phases, an intensive communication strategy on end-of-life practice was implemented based on the framework developed at the International Delphi Conference. The following data were recorded for all participating nurses: age, gender, marital status, years of practice since certification, and years of critical care experience; the following data on ICU status were also collected from the electronic system: total number of patients, length of ICU stay, ICU mortality rate, in-hospital mortality rate, ICU admission APACHE-II score, SOFA score at ICU admission, and medical costs at ICU admission. Continuous variables without normal distribution are shown as median and interquartile range. Categorical data were summarized numerically or as percentages. In univariate analyses, Mann-Whitney's U test was used to compare continuous variables and Fisher's exact test to compare categorical variables. Data were assumed to be missing at random, and no imputation or interpolation of missing values was performed. Statistical tests were two-tailed and statistical significance was set at p<0.05. All statistical analyses were performed using EZR (R Foundation for Statistical Computing, Vienna, Austria), a graphical user interface for R. The study was approved by the Maebashi Red Cross Hospital Ethics Committee (ID: 2022-47), which waived the requirement for informed consent from patients and their relatives, given the retrospective and observational nature of the study.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses working in our ICU

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The Japanese Quality of Dying and Death (QODD) in ICU | Approximately one month
  The Japanese Quality of Dying and Death (QODD) in ICU consists of six items, each of which is rated on a scale of 0 to 10, with higher scores indicating higher quality of death. It is based on the U.S. Intensive Care Unit version of the Quality of Dying and Death (ICU-QODD) and was adapted to Japanese culture, and its validation has been confirmed.
The Japanese Burnout Scale | Approximately one month
  The Japanese Burnout Scale consists of 17 items, each with a score of 1-5, with higher scores indicating stronger burnout symptoms. It assesses subjects' burnout symptoms and is based on the Massachusetts Burnout Inventory. The scale was developed for the Japanese culture based on the Massluck Burnout Inventory, and its validation has been verified.

SECONDARY OUTCOMES:
The medical costs in ICU | Approximately one month
  Calculated for the total medical costs incurred in the ICU
The length of ICU stay | Approximately one month
  Calculated as the average number of days per stay per patient
Mortality at ICU | Approximately one month

CONTACTS AND LOCATIONS:
Locations (1):
- Maebashi Redcross hospital, Maebashi, Gunma, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quenot JP, Rigaud JP, Prin S, Barbar S, Pavon A, Hamet M, Jacquiot N, Blettery B, Herve C, Charles PE, Moutel G. Suffering among carers working in critical care can be reduced by an intensive communication strategy on end-of-life practices. Intensive Care Med. 2012 Jan;38(1):55-61. doi: 10.1007/s00134-011-2413-z. Epub 2011 Nov 30. PMID 22127481
- [Background] Kerckhoffs MC, Senekal J, van Dijk D, Artigas A, Butler J, Michalsen A, van Mol MMC, Moreno R, Pais da Silva F, Picetti E, Povoa P, Robertsen A, van Delden JJM. Framework to Support the Process of Decision-Making on Life-Sustaining Treatments in the ICU: Results of a Delphi Study. Crit Care Med. 2020 May;48(5):645-653. doi: 10.1097/CCM.0000000000004221. PMID 32310619